CLINICAL TRIAL: NCT06308367
Title: The Effect of Betaine in Refractory Syringomyelia（RS）
Brief Title: The Therapeutic Effect of Betaine in Syringomyelia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XWTEBS
Record Dates: First submitted 2024-02-17; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Syringomyelia
MeSH Terms: conditions — Syringomyelia | interventions — Betaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- betaine (Experimental): oral betaine
  Interventions: Drug: Betaine
- placebo (Placebo Comparator): rice-flour as a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Betaine — 50mg/kg for 12 weeks
  Arms: betaine
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
Purpose: This clinical trial aims to evaluate the indications, therapeutic effects and side effects of betaine in refractory syringomyelia.

Primary outcome measure: The primary endpoint is the change of ASIA at week 12. The clinical efficacy is defined as ASIA increase ≥ 1 at week 12, as compared with that before betaine usage.

DETAILED DESCRIPTION:
The pathogenesis of syringomyelia is poorly understood and duraplasty or shunting is not always effective. Although it is generally thought that syringomyelia is simply an accumulation of CSF from the subarachnoid space, the pathogenesis is likely to be more complex and may involve cellular and molecular processes.

The investigators supposed that betaine might play a key role in the pathogenesis of syringomyelia, especially post-traumatic syringomyelia(PTS), and that betaine, as an Osmotic homeostasis-related drug, would protect Osmotic homeostasis in syringomyelia.

Primary objectives: This clinical trial aims to evaluate the indications, therapeutic effects and safety of betaine in refractory syringomyelia.

ELIGIBILITY:
Inclusion Criteria:

* Contraindication to duraplasty and shunting treatment due to history or high risk of severe adverse effects,
* non-effective response to duraplasty and shunting treatment in 12 months prior to study entry.
* Estimated life expectancy must be greater than 12 months.
* Ability to understand and willingness to sign a written informed consent document, or constant caregivers who well understand and willingness to sign a written informed consent document.
* Must be able to swallow tablets

Exclusion Criteria:

* Participants have a cardiometabolic disease for which they take prescribed medications
* Evidence of tumor metastasis, recurrence, or invasion;
* History of psychiatric diseases ;
* History of seizures;
* History of arteriosclerotic cardiovascular diseases (ASCVD), e.g. stroke, myocardial infaction, unstable angina, within 6 months;
* New York Heart Association Grade II or greater congestive heart failure;
* Serious and inadequately controlled cardiac arrhythmia;
* Significant vascular disease, e.g. moderate or severe carotid stenosis, aortic aneurysm, -history of aortic dissection;
* Severe infection;
* History of allergy to relevant drugs;
* Pregnancy, lactation, or fertility program in the following 12 months;
* History or current diagnosis of peripheral nerve disease;
* Abnormal in liver and renal function;
* Active tuberculosis;
* Transplanted organs;
* Human immunodeficiency virus;
* Participation in other experimental studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
ASIA Score | 1 day before and 3 days, 3 months, after drug treatment
  American Spinal Injury Association(ASIA) Score for evaluating the spinal cord function， degree of the spinal cord function, motor1-100, sensory 1-224, higher scores mean a better outcome

SECONDARY OUTCOMES:
syringomyelia remission | 1 day before and 3 days, 3 months, after drug treatment
  syringomyelia remission is defined as ≥ 25% reduction in syringomyelia volume on T2 images at week 12, as compared with that before thalidomide usage
Electrophysiology results | 1 day before and 3 days, 3 months, after drug treatment
  electromyography and evoked potential; Change of N9-13 From Baseline in Electrophysiology at postoperation
Visual Analog Scale (VAS) | 1 day before and 3 days, 3 months, after drug treatment
  degree of the pain, 1-10, higher scores mean a worse outcome
Klekamp and Sammi syringomyelia scale | 1 day before and 3 days, 3 months, after drug treatment
  for evaluating the spinal cord function, higher scores mean a better outcome
modified Japanese Orthopaedic Association Scores (mJOA) | 1 day before and 3 days, 3 months, after drug treatment
  Motor function， sensory， bladder function；for evaluating the spinal cord function；0-17， higher scores mean a better outcome
xuanwu syringomyelia scale | 3 days, 3 months, after drug treatment
  for evaluating the spinal cord function, for evaluating the spinal cord function；0-18， higher scores mean a worse outcome
Incidence of complications | 3 days, 3 months, after drug treatment
  Incidence of complications

CONTACTS AND LOCATIONS:
Locations (1):
- Fengzeng Jian, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guan J, Yuan C, Yao Q, Du Y, Fang Z, Zhang L, Jia S, Zhang C, Liu Z, Wang K, Duan W, Wang Z, Wang X, Wu H, Chen Z, Jian F. A novel scoring system for assessing adult syringomyelia associated with CM I treatment outcomes. Acta Neurol Belg. 2023 Jun;123(3):807-814. doi: 10.1007/s13760-023-02264-4. Epub 2023 Apr 12. PMID 37046133
- [Background] Mohrman AE, Farrag M, Huang H, Ossowski S, Haft S, Shriver LP, Leipzig ND. Spinal Cord Transcriptomic and Metabolomic Analysis after Excitotoxic Injection Injury Model of Syringomyelia. J Neurotrauma. 2017 Feb;34(3):720-733. doi: 10.1089/neu.2015.4341. Epub 2016 Oct 13. PMID 27736311
- [Background] He R, Zhang H, Kang L, Li H, Shen M, Zhang Y, Mo R, Liu Y, Song J, Chen Z, Liu Y, Jin Y, Li M, Dong H, Zheng H, Li D, Qin J, Zhang H, Huang M, Liang D, Tian Y, Yao H, Yang Y. Analysis of 70 patients with hydrocephalus due to cobalamin C deficiency. Neurology. 2020 Dec 8;95(23):e3129-e3137. doi: 10.1212/WNL.0000000000010912. Epub 2020 Sep 17. PMID 32943488
- [Result] Hemley SJ, Bilston LE, Cheng S, Stoodley MA. Aquaporin-4 expression and blood-spinal cord barrier permeability in canalicular syringomyelia. J Neurosurg Spine. 2012 Dec;17(6):602-12. doi: 10.3171/2012.9.SPINE1265. Epub 2012 Oct 19. PMID 23082850
- [Result] Yuan C, Xia P, Duan W, Wang J, Guan J, Du Y, Zhang C, Liu Z, Wang K, Wang Z, Wang X, Wu H, Chen Z, Jian F. Long-Term Impairment of the Blood-Spinal Cord Barrier in Patients With Post-Traumatic Syringomyelia and its Effect on Prognosis. Spine (Phila Pa 1976). 2024 Mar 15;49(6):E62-E71. doi: 10.1097/BRS.0000000000004884. Epub 2023 Nov 28. PMID 38014747
- [Result] Heiss JD. Cerebrospinal Fluid Hydrodynamics in Chiari I Malformation and Syringomyelia: Modeling Pathophysiology. Neurosurg Clin N Am. 2023 Jan;34(1):81-90. doi: 10.1016/j.nec.2022.08.007. Epub 2022 Nov 3. PMID 36424067
- [Result] Guan J, Yuan C, Zhang C, Ma L, Yao Q, Cheng L, Liu Z, Wang K, Duan W, Wang X, Wu H, Chen Z, Jian F. Intradural Pathology Causing Cerebrospinal Fluid Obstruction in Syringomyelia and Effectiveness of Foramen Magnum and Foramen of Magendie Dredging Treatment. World Neurosurg. 2020 Dec;144:e178-e188. doi: 10.1016/j.wneu.2020.08.068. Epub 2020 Aug 15. PMID 32805463
- [Result] Liu S, Ma L, Qi B, Li Q, Chen Z, Jian F. Suppression of TGFbetaR-Smad3 pathway alleviates the syrinx induced by syringomyelia. Cell Biosci. 2023 May 29;13(1):98. doi: 10.1186/s13578-023-01048-w. PMID 37248485